CLINICAL TRIAL: NCT05688657
Title: Clinical Evaluation of Clariti Monthly Toric and Clariti 1 Day Toric
Brief Title: Clinical Evaluation of Two Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-137
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: All participants received Lens A and then Lens B in fixed-sequence order.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (Experimental): All participants wore Lens A for 15 minutes (Period 1)
  Interventions: Device: Lens A
- Lens B (Experimental): All participants wore Lens B for 15 minutes (Period 2)
  Interventions: Device: Lens B

INTERVENTIONS:
Device: Lens A — Monthly Replacement Toric Silicone Hydrogel Contact Lens 15 minutes of daily wear
  Arms: Lens A
Device: Lens B — Daily Disposable Toric Silicone Hydrogel Contact Lens 15 minutes of daily wear
  Arms: Lens B

SUMMARY:
The study objective was to compare short-term clinical performance data of two toric contact lenses.

DETAILED DESCRIPTION:
The aim of this non-dispensing fitting study was to evaluate the short-term clinical performance of a monthly toric contact lens when compared to a daily disposable toric contact lens after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Is not a habitual wearer of either study lens
* Has a contact lens spherical prescription between +4.00 to -9.00 (inclusive) best corrected visual acuity of 20/30 or better in either eye
* Have contact lens prescription of no less than -0.75D of astigmatism and no more than -2.25 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.50 D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:
* Pathological dry eye or associated findings
* Pterygium, pinguecula, or corneal scars within the visual axis
* Neovascularization > 0.75 mm in from of the limbus
* Giant papillary conjunctivitis (GCP) worse than grade 1
* Anterior uveitis or iritis (past or present)
* Seborrheic eczema, Seborrheic conjunctivitis
* History of corneal ulcers or fungal infections
* Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén V Guerrero, MSc., FIACLE, Principal Investigator — Dr. Ruben Velazquez Private Practice
Locations (1):
- Dr. Ruben Velazquez Private Practice, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-two participants were screened. All participants wore Lens A for first 15 minutes and then wore Lens B for 15 minutes.
  All the participants who were in the study were included in the analysis. (n=42)
Groups:
- Lens A: All participants wore Lens A for 15 minutes. (Period 1)
- Lens B: All participants wore Lens B for 15 minutes. (Period 2)
Period: Period 1: Lens A (15 Minutes)
Arm/Group | Lens A | Lens B
Started | 42 | 0 (All participants received Lens A in Period 1.)
Completed | 42 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B (15 Minutes)
Arm/Group | Lens A | Lens B
Started | 0 (All participants received Lens B in Period 2.) | 42
Completed | 0 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  Lens A: <=18 years | 0
  Lens A: Between 18 and 65 years | 42
  Lens A: >=65 years | 0
  Lens B: <=18 years | 0
  Lens B: Between 18 and 65 years | 42
  Lens B: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Handling Ratings on Insertion
Description: Subjective handling ratings on insertion will be measured on a scale from 0-100, where (0= extremely uncomfortable) and 100 = better performance
Time Frame: At insertion
Population: [Not Specified]
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants that received Lens A.
- Lens B: Participants that received Lens B.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 42 | 42
units on a scale | 92.0 (13.1) | 93.7 (9.2)

ADVERSE EVENTS:
Time Frame: From dispense up to 15mins on each lens type.
Description: [Not specified]
Groups:
- Lens A: Participants wore Lens A for 15mins.
- Lens B: Participants wore Lens B for 15mins.
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT05688657/Prot_SAP_000.pdf